CLINICAL TRIAL: NCT02125266
Title: A Prospective, Multi-Center, Randomized, Controlled Clinical Trial Designed to Evaluate the Safety and Preliminary Efficacy of V404 PDS in Chronic Noninfectious Uveitis
Brief Title: Safety and Preliminary Efficacy Study of V404 PDS in Uveitis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to unacceptable frequency of drug related adverse events
Sponsor: Forsight Vision4 (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V4041
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Uveitis, Posterior; Uveitis, Intermediate
MeSH Terms: conditions — Uveitis, Posterior; Uveitis, Intermediate | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose V404 PDS (Experimental): Sustained intravitreal delivery of methotrexate (0.6 mg)
  Interventions: Drug: V404
- High Dose V404 PDS (Experimental): Sustained intravitreal delivery of methotrexate (2.3 mg)
  Interventions: Drug: V404

INTERVENTIONS:
Drug: V404 — Sustained Release
  Other Names: Methotrexate

SUMMARY:
This study is intended to evaluate the safety of V404 PDS in patients with chronic non-infectious uveitis. Secondarily, the study will evaluate whether V404 PDS can provide clinically measurable benefit over an extended period of time in patients with chronic non-infectious uveitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Confirmed diagnosis of active uveitis
* Sufficient lens/media clarity
* Meet best-corrected visual acuity criteria
* Willing and able to use contraception

Exclusion Criteria:

* Pregnant, breast feeding
* Uncontrolled glaucoma
* Intraocular surgery or periocular/intraocular injections within 6 weeks
* Periocular or intraocular steroid within 3 months
* Prior vitrectomy
* Prior corneal transplant
* Prior fluocinolone implant
* Allergy or sensitivity to study drug
* Participation in other trial within 30 days
* Abnormal liver function
* History of positive serum tuberculosis test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | 6 months

SECONDARY OUTCOMES:
Change in vitreous haze score | Baseline, 6 Months

OTHER OUTCOMES:
Change in macular thickness by ocular coherence tomography | Baseline, 6 Months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Golden, Colorado
  - Atlanta, Georgia
  - Omaha, Nebraska
  - Cleveland, Ohio
  - Arlington, Texas

IPD SHARING:
Plan to Share IPD: No